CLINICAL TRIAL: NCT04925375
Title: Abatacept for the Treatment of Common Variable Immunodeficiency With Interstitial Lung Disease
Acronym: ABCVILD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0876; R01FD007267 (FDA)
Record Dates: First submitted 2021-05-11; First posted 2021-06-14 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Interstitial Lung Disease; Common Variable Immunodeficiency
MeSH Terms: conditions — Lung Diseases, Interstitial; Common Variable Immunodeficiency | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: Randomized, blinded/placebo-controlled clinical trial in pediatric and adult subjects ≥50 kg (cohort 1), with an additional cohort (#2) of pediatric subjects <50 kg tested as a single arm, receiving open-label abatacept
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abatacept (Experimental): Pediatric subjects weighing <50 kg will be placed in an single arm with abatacept with dosing based on weight. Pediatric subjects weighing ≥50kg and adult subjects will enter a double blinded, randomization in a 1:2 ratio of subjects to the abatacept treatment group (arm 1) or to the placebo group (arm 2) treated weekly through month 6. After month 6, all subjects will begin receiving abatacept weekly.
  Pediatric dosing:
  Abatacept subcutaneous every week:
  10-25 kg: 50 mg; 25-50 kg: 87.5 mg; >50 kg: 125 mg
  Adult dosing:
  Abatacept: 125 mg subcutaneous every week
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): Pediatric subjects weighing ≥50kg and adult subjects will enter a double blinded, randomization in a 1:2 ratio of subjects to the abatacept treatment group (arm 1) or to the placebo group (arm 2) treated weekly through month 6. The composition of the placebo is the same as the active study drug without the abatacept. To maintain the blind, injection volumes will be the same as the active treatment. After month 6, all subjects will begin receiving abatacept weekly.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Abatacept — Abatacept is a selective costimulation modulator, inhibiting T lymphocyte activation by binding to CD80 and CD86, thereby blocking interaction with CD28. Orencia solution supplied in a prefilled syringe should be refrigerated at 2C to 8C (36F to 46F). Orencia should not be used beyond the expiration date on the prefilled syringe. The product should be protected from light by storing in the original package until time of use. The prefilled syringe should not be frozen.
  Other Names: Orencia
  Arms: Abatacept
Other: Placebo — The composition of the placebo for Orencia is the same as the active study drug without the abatacept. The placebo will be packaged and labeled as described above for the Orencia prefilled syringes. To maintain the blind, injection volumes will be the same as the active treatment.
  Arms: Placebo

SUMMARY:
There is no standard of care therapy for patients with granulomatous-lymphocytic interstitial lung disease (GLILD) seen in common variable immunodeficiency (CVID). Abatacept has recently looked promising for the treatment of patients with complex CVID. This study is a multi-site, phase II, randomized, blinded/placebo-controlled clinical trial in pediatric and adult subjects to determine the efficacy of abatacept compared to placebo for treatment of subjects with GLILD in the context of CVID.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
There is no standard of care therapy for patients with granulomatous-lymphocytic interstitial lung disease (GLILD) seen in common variable immunodeficiency (CVID). Abatacept is a recombinant, human fusion protein of cytotoxic T lymphocyte-associated protein 4 (CTLA-4) and human IgG1 that blocks T cell activation by binding to CD80 and CD86, thereby blocking CD28 engagement- the "second signal" needed for T cell activation. Abatacept has recently looked promising for the treatment of patients with complex CVID.

This study is a multi-site, phase II, randomized, blinded/placebo-controlled clinical trial in pediatric subjects ≥50 kg and adult subjects (cohort 1), with an additional cohort (#2) of pediatric subjects <50 kg tested as a single arm, receiving open-label abatacept. Cohort 1 utilizes a 'delayed-start' design to obtain maximum statistical power from this cohort. Cohort 2 will be open label due to the lack of a suitable placebo for pediatric dose abatacept syringes. A total of 21-30 evaluable subjects will be treated in cohort 1 and 8 evaluable subjects in cohort 2.

Following the initial 12 months of treatment, patients will have the option of continuing abatacept for up to 3 years. Patients will have the option of continuing abatacept any time after the initial 12 months of treatment (does not have to be immediately). A separate consent form will be utilized to document a patient's decision to continue. Abatacept will be provided by BMS. Patients who decide to continue abatacept will be monitored for safety, including infections, approximately every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CVID according to the international consensus document (ICON)

   1. Age 4 years or above
   2. Serum IgG at least 2 standard deviations below the age adjusted normal
   3. Decreased serum IgA and/or serum IgM
   4. Abnormal specific antibody response to immunization
   5. Exclusion of secondary immunodeficiency
2. On replacement immunoglobulin for at least 6 months and willing to maintain throughout study
3. Granulomatous-lymphocytic interstitial lung disease with a lymphocytic component diagnosed by lung biopsy prior to study entry, wedge biopsy preferred.
4. Persistence or worsening of interstitial lung disease measured on serial CT imaging of the lung at least 6 months apart, with the latest assessment within 3 months of study entry.
5. Signed written informed consent
6. Willing to allow storage of biological specimens for future use in medical research.
7. Female subjects of childbearing potential must agree to an effective form of birth control such as hormone based contraceptive, intrauterine device, condoms/barrier, surgically sterile partner, or abstinence.
8. Fertile, non-vasectomized males with a female partner of childbearing potential should use condoms throughout the study and for 3 months after the last dose

Exclusion Criteria:

1. History of hypersensitivity to abatacept or any of its components
2. Has received any lymphocyte depleting agents including anti-CD20 monoclonal antibodies, alemtuzumab, ATG in the preceding 6 months
3. Has received abatacept, cyclophosphamide, tumor necrosis factor inhibitors, or pulse steroids (defined as >15mg/kg/day of methylprednisone or corticosteroid equivalent) within the past 3 months
4. Have started or increased any of the following immune modulating drugs within 3 months of enrolling and 3 months from initial CT chest: azathioprine, cyclosporine, tacrolimus, mercaptopurine, methotrexate, mycophenolate mofetil, or sirolimus
5. History of HIV infection (positive PCR)
6. Chronic untreated hepatitis B or C (positive PCR)
7. Active tuberculosis (TB) by positive QuantiFERON gold. If history of latent TB, then must supply evidence of completing treatment.
8. Persistent Epstein-Barr Virus (EBV) load ≥ 1,000 units/mL blood checked twice at least 1 month apart
9. Other uncontrolled infections
10. Live vaccine given within 6 weeks of the start of the trial
11. Malignancy or treated for malignancy within the past year
12. Currently pregnant or breast feeding
13. Life expectancy less than 1 month
14. Subjects unwilling to self-administer or have a parent/caregiver self-administer subcutaneous injections at home
15. Other conditions that the investigators feel contraindicate participation in the study

Inclusion criteria for Extended Treatment Plan:

* Patients must have completed the abatacept for the treatment of Interstitial Lung Disease in Common Variable Immunodeficiency (ABCVILD) trial
* Patients must have demonstrated positive response to abatacept.
* Patients must provide informed consent to participate in the Extended Treatment Plan.

Exclusion criteria for Extended Treatment Plan:

• Patients who experienced SAEs during the original trial, and such SAEs were determined as related to treatment, or patients who in the opinion of the investigator would not benefit from the extended treatment option.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
High Resolution CT Scan of the chest (HRCT) | 6 months
  Proportion of subjects achieving a significant response (defined as >30 percent change in lung tissue disease burden by GLILD) on HRCT after 6 months of abatacept therapy.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 6 months, 12 months
  Forced vital capacity (FVC)
Forced expiratory volume (FEV) | 6 months, 12 months
  Forced expiratory volume (FEV)
Diffusion capacity of carbon monoxide (DLCo) | 6 months, 12 months
  Diffusion capacity of carbon monoxide (DLCo)
Incidence | 6 months, 12 months
  Incidence of new onset autoimmune/inflammatory diseases while on abatacept or placebo
Resolution | 6 months, 12 months
  Resolution of existing autoimmune/inflammatory diseases while on abatacept or placebo
Change in Short Form-36 scores | 6 months, 12 months
  Short Form-36: scoring ranges from 0-100 where a higher score denotes better health
Change in PedsQL (Pediatric Quality of Life) Generic Core scores | 6 months, 12 months
  PedsQL Generic Core Scales: items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL. Range of 0-2300 for ages above 4, range of 0-2100 for 4 years old
Change in King's Interstitial Lung Disease scores | 6 months, 12 months
  King's Interstitial Lung Disease: scoring ranges from 0-100 where a higher score denotes better health
Steroid usage | 6months, 12 months
  Cumulative number of steroids used after 6 months and 12 months
Survival | 6 months, 12 months
  Survival at 12 months
Pediatric growth - change in height | 6 months, 12 months
  Change in height at 6 and 12 months.
Pediatric growth - change in weight | 6 months, 12 months
  Change in weight at 6 and 12 months.
Additional Immune Agents | 6 months, 12 months
  Rate of discontinuation of additional immune agents while on study agent
Adverse Events/Serious Adverse Events | 6 months, 12 months
  Incidence of adverse events and severe adverse events, compared to placebo
Dropout rate | 6 months, 12 months
  Study dropout rate
Incidence of concurrent infections | 6 months, 12 months
  Incidence of concurrent infections while on study
Treatment of concurrent infections | 6 months, 12 months
  Number of infections per patient which require treatment with antibiotics
Complications of concurrent infections | 6 months, 12 months
  Complications of concurrent infections while on study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jordan, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - University of South Florida, Tampa, Florida
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No